CLINICAL TRIAL: NCT06139263
Title: The Effect of Vibration Therapy on Pain, Functionality and Proprioception in İndividuals With Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-1701
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cervical Disc Herniation; Vibration Therapy; Pain; Functionality; Proprioception
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): All individuals participating in the study will receive a conventional treatment program 4 days a week. In the conventional treatment program, heat will be applied to the neck area for 20 minutes and TENS (100 Hz) will be applied to the painful area. Additionally, patients will be given joint range of motion (ROM) exercises under the supervision of a physiotherapist. Patients will be asked to perform ROM exercises in 2 sets of 10 repetitions, holding for 2 seconds at the end point in all directions. As a strengthening exercise, isometric exercises will be given in the flexion extension, right and left lateral flexion directions by waiting for 6 seconds at the end point. Isometric exercises will be performed in 2 sets of 10 repetitions with 1 minute rest between sets.
  Interventions: Other: conventional treatment program
- Vibration Group (Experimental): Vibration application will be applied to the individuals in this group in addition to conventional methods. Vibration application will be applied to the trapezius, levator scapula and cervical paravertebral muscles with a percussion massage gun (Compex Fix 2.0) along the origo-insersio line for 3 minutes for each muscle group. Vibration application will be made with the soft head of the percussion massage gun. Vibration therapy will be applied 3 days a week for 3 weeks.
  Interventions: Device: a percussion massage gun (Compex Fix 2.0); Other: conventional treatment program

INTERVENTIONS:
Device: a percussion massage gun (Compex Fix 2.0) — Vibration application will be applied to the individuals in this group in addition to conventional methods. Vibration application will be applied to the trapezius, levator scapula and cervical paravertebral muscles with a percussion massage gun (Compex Fix 2.0) along the origo-insersio line for 3 minutes for each muscle group. Vibration application will be made with the soft head of the percussion massage gun. Vibration therapy will be applied 3 days a week for 3 weeks.
  Arms: Vibration Group
Other: conventional treatment program — In the conventional treatment program, heat will be applied to the neck area for 20 minutes and TENS (100 Hz) will be applied to the painful area. Additionally, patients will be given joint range of motion (ROM) exercises under the supervision of a physiotherapist. Patients will be asked to perform ROM exercises in 2 sets of 10 repetitions, holding for 2 seconds at the end point in all directions. As a strengthening exercise, isometric exercises will be given in the flexion extension, right and left lateral flexion directions by waiting for 6 seconds at the end point. Isometric exercises will be performed in 2 sets of 10 repetitions with 1 minute rest between sets.

SUMMARY:
This study aimed to examine the effects of vibration applied at different frequencies with a percussion massage gun on joint range of motion, pain, functionality and kinesiophobia in individuals with cervical disc herniation.All individuals participating in the study will receive a conventional treatment program. In the conventional treatment program, heat will be applied to the neck area for 20 minutes and TENS (100 Hz) will be applied to the painful area. Additionally, patients will be given joint range of motion (ROM) exercises under the supervision of a physiotherapist.

Vibration Group Vibration application will be applied to the individuals in this group in addition to conventional methods. Vibration application will be applied to the trapezius, levator scapula and cervical paravertebral muscles with a percussion massage gun (Compex Fix 2.0) along the origo-insersio line for 3 minutes for each muscle group. Vibration application will be made with the soft head of the percussion massage gun. Vibration therapy will be applied 3 days a week for 3 weeks.

DETAILED DESCRIPTION:
This study aimed to examine the effects of vibration applied at different frequencies with a percussion massage gun on joint range of motion, pain, functionality and kinesiophobia in individuals with cervical disc herniation.All individuals participating in the study will receive a conventional treatment program 4 days a week. In the conventional treatment program, heat will be applied to the neck area for 20 minutes and TENS (100 Hz) will be applied to the painful area. Additionally, patients will be given joint range of motion (ROM) exercises under the supervision of a physiotherapist. Patients will be asked to perform ROM exercises in 2 sets of 10 repetitions, holding for 2 seconds at the end point in all directions. As a strengthening exercise, isometric exercises will be given in the flexion extension, right and left lateral flexion directions by waiting for 6 seconds at the end point. Isometric exercises will be performed in 2 sets of 10 repetitions with 1 minute rest between sets.

Vibration Group Vibration application will be applied to the individuals in this group in addition to conventional methods. Vibration application will be applied to the trapezius, levator scapula and cervical paravertebral muscles with a percussion massage gun (Compex Fix 2.0) along the origo-insersio line for 3 minutes for each muscle group. Vibration application will be made with the soft head of the percussion massage gun. Vibration therapy will be applied 3 days a week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with cervical disc herniation,
* Having complained of neck pain for at least 3 weeks,
* Individuals with limited neck joint range of motion.

Exclusion Criteria:

* Those who have another orthopedic or neurological disorder in addition to their neck problem,
* Having a history of previous trauma in the neck area,
* Included in the physiotherapy program in the last 6 months,
* Individuals who cannot tolerate vibration application.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of Joint Position Sense | 10 minutes
  Patients' joint position sense will be evaluated with the Laser Cursor Assisted Angle Repetition Test (LI-YATT).

SECONDARY OUTCOMES:
Neck Disability Index | 10 minutes
  The Neck Disability Index (NDI) scale will be used to evaluate neck disability. NDI is an easy-to-apply, reliable, and validated index used by Vernon and Mior to measure pain and limitations in daily living activities caused by neck pathologies. This index consists of 10 parts with headings such as severity of pain, lifting loads, reading, headache, personal care, business life, concentration, sleep, recreational activities and driving, and there are 6 answers for each heading ranging from 0 to 5 points. 0 indicates that there is no pain or any functional limitation, while 5 indicates that the most pain and limitation is present.
Visual Analogue Scale | 5 minutes
  Visual Analogue Scale (VAS) will be used to evaluate the pain intensity of patients. VAS consists of a 10 cm long horizontal line. '0' represents no pain, '10' represents unbearable pain. During our evaluation, patients will be asked to mark the level of pain they feel on this chart, and the distance to the starting point will be measured and recorded with the ruler.
Kinesiophobia | 10 minutes
  The patients' kinesiophobia will be evaluated with the Tampa Kinesiophobia Scale (TKÖ). This scale was developed by Kori et al. to evaluate patients' fear of movement. It is a 17-question scale prepared by A.Ş. in 1990 and has Turkish validity and reliability. The scoring of this 4-point Likert type scale is; "strongly disagree" is 1, "disagree" is 2, 26 "agree" is 3, "strongly agree" is 4. A total score is calculated after reversing the 4th, 8th, 12th and 16th items. The person receives a total score between 17-68. The higher the score a person gets on the scale, the higher the degree of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, Phd, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No